CLINICAL TRIAL: NCT05520866
Title: PrehabPal: A Digital Tool to Help Frail Elders Prepare for Cancer Surgery
Brief Title: PrehabPal: A Digital Tool to Help Older Adults Prepare for Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Emerson Collective (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 228013; 22-37253 (Other: University of California, San Francisco); NCI-2023-02952 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Colon Cancer
Keywords: Web app; Older Adult; Prehabilitation
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrehabPal Web app (Experimental): Web app based initial geriatric assessment will be given followed by daily tailored prehabilitation activities in the domains of exercise, nutrition, anxiety reduction, home preparation, and advanced care planning. Each participant is paired with a central health coach who monitors engagement and provides support through the Web app portal.
  Interventions: Behavioral: PrehabPal
- Written Surgery Prehabilitation Instructions (No Intervention): Participants will be provided paper-based prehabilitation instructions that include information about exercise, nutrition, anxiety reduction, home preparation, and advanced care planning. A paper diary is provided to record any prehabilitation activities.

INTERVENTIONS:
Behavioral: PrehabPal — Web based application
  Arms: PrehabPal Web app

SUMMARY:
This is a multi-center, randomized trial investigating the use of PrehabPal web app versus a written surgery prehabilitation instructions among individuals aged 65 years and older preparing for colon cancer surgery. PrehabPal is a web app designed with, and for, older adults preparing for surgery at University of California, San Francisco (UCSF). This app has the potential to fill a crucial clinical gap for older cancer patients by designing an individualized prehabilitation program and providing prehabilitation coaching.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effectiveness of PrehabPal in delivering prehabilitation and improving outcomes for elders who undergo colorectal cancer surgery.

SECONDARY OBJECTIVES:

I. Determine the impact of PrehabPal on surgical outcomes and functional recovery compared to standard written surgery prehabilitation materials.

OUTLINE:

Participants will be randomly assigned to 1 of 2 conditions. Study participation will continue for up to 12 weeks, with intervention 7-21 days before surgery and a follow-up visit 8 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >=65 years of age at time of evaluation for colorectal cancer resection.
2. Documentation of a colorectal diagnosis as evidenced by the following criteria:

   a. Biopsy proven colorectal cancer or unresectable neoplastic polyp.
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
4. Self-reported access to the Internet.
5. Participant has at least seven days prior to surgery date to optimize for surgery.
6. English language proficient.

Exclusion Criteria:

1. No English language proficiency.
2. No Internet access.
3. Documented diagnosis of dementia or Alzheimer's disease.
4. Surgery scheduled within 7-days.
5. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of days before surgery engaged in prehabilitation | Up to 14 days
  The proportion of days before surgery engaged in prehabilitation between subjects randomized to the PrehabPal Web App and written prehabilitation materials using logistic regression. Since sites may not balance, all relevant sociodemographic and clinical characteristics of the subjects may be included in the models which will include other factors that are not balanced between the sites.

SECONDARY OUTCOMES:
Proportion of participants with reported Surgical Complications | 30 days following surgery
  Incidence of reported adverse events 30 days after surgery will be classified according to the Clavien-Dindo complications index.
Median Length of Stay (LOS) | Post procedure until discharge, approximately 2 days
  The median time from surgery until discharge from hospital will be reported.
Readmission Rate | 30 days following surgery
  The proportion of participants who were re-admitted to the hospital within 30 days of surgery will be reported.
Change in Mean score on the SF-36 | Up to 8 weeks
  Short Form 36 (SF-36) Health Survey: includes 36 items or questions that assess functional health and well-being from the perspective of the patient. The items contribute to eight health domains of physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. The eight domains all contribute to physical component summary (PCS) and mental component summary (MCS) scores Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability. The calculated composite scores of the Physical Component Scale (PCS) and the Mental Component Scale (MCS) scores of the SF-36 will be measured at baseline and 8 weeks post surgery

OTHER OUTCOMES:
Median Satisfaction Scores | 8 weeks post-surgery
  Patient-participant reported satisfaction with the PrehabPal web app and the paper-mode activities diary will be measured via a survey created by the investigators in REDCap.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Finlayson, MD, MS, FACS, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carli F, Bousquet-Dion G, Awasthi R, Elsherbini N, Liberman S, Boutros M, Stein B, Charlebois P, Ghitulescu G, Morin N, Jagoe T, Scheede-Bergdahl C, Minnella EM, Fiore JF Jr. Effect of Multimodal Prehabilitation vs Postoperative Rehabilitation on 30-Day Postoperative Complications for Frail Patients Undergoing Resection of Colorectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Mar 1;155(3):233-242. doi: 10.1001/jamasurg.2019.5474. PMID 31968063
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Derived] Ogomori K, Broering J, Rogine C, Kin C, Chang GJ, Finlayson E. Evaluating a digital prehabilitation tool in patients with colorectal surgery: protocol for a multisite randomised controlled trial. BMJ Open. 2025 Feb 18;15(2):e088001. doi: 10.1136/bmjopen-2024-088001. PMID 39965940